CLINICAL TRIAL: NCT07216235
Title: A Phase 3b/4, Multicenter, Parallel-Group, Double-Blind, Placebo Controlled, Two-Arm, Long-Term Study to Evaluate the Safety and Efficacy of Saroglitazar Magnesium on Clinical Outcomes in Participants With Primary Biliary Cholangitis (PBC)
Brief Title: Long-Term Study to Evaluate the Safety and Efficacy in Participants With Primary Biliary Cholangitis of Saroglitazar Magnesium-V on Clinical Outcomes
Acronym: EPICS-V
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SARO.23.001
Record Dates: First submitted 2025-10-05; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Primary Biliary Cholangitis
Keywords: Saroglitazar Magnesium; Primary Biliary Cholangitis; PBC; clinical outcome
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — saroglitazar

STUDY DESIGN:
Intervention Model Description: Phase 3b/4, Multicenter, Parallel-Group, Double-Blind, Placebo-Controlled, safety and efficacy study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saroglitazar 1 mg (Experimental): Saroglitazar magnesium 1 mg, once daily, orally each morning before breakfast
  Interventions: Drug: Saroglitazar magnesium 1 mg
- Placebo (Placebo Comparator): Matching placebo once daily orally each morning before breakfast
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saroglitazar magnesium 1 mg — Saroglitazar magnesium 1 mg once daily, orally each morning before breakfast
  Arms: Saroglitazar 1 mg
Drug: Placebo — Matching Placebo once daily, orally each morning before breakfast
  Arms: Placebo

SUMMARY:
Long-Term Study to Evaluate the Safety and Efficacy in Participants with Primary Biliary Cholangitis of Saroglitazar Magnesium-V on Clinical Outcomes (EPICS-V)

DETAILED DESCRIPTION:
A Phase 3b/4, Multicenter, Parallel Group, Double Blind, Placebo Controlled, Two Arm, Long Term Study to Evaluate the Safety and Efficacy of Saroglitazar Magnesium on Clinical Outcomes in Participants with Primary Biliary Cholangitis (PBC)

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following criteria to be enrolled in this study:

1. Is capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with protocol requirements
2. Is an adult male or female, must be ≥18 years of age at the time of signing informed consent
3. Is receiving ursodeoxycholic acid (UDCA) for ≥12 months with a stable dose for ≥6 months prior to screening,and expected to remain on a stable dose during the study period OR Is unable to tolerate UDCA and did not receive UDCA in the past 3 months prior to screening
4. Has a history of confirmed PBC diagnosis, as demonstrated by the presence of ≥2 of the following 3 diagnostic factors:

   i. A history of elevated ALP levels for ≥6 months prior to screening ii. Positive antimitochondrial antibodies (AMA) titer OR if AMA is negative, then positive PBC-specific antibodies iii. Liver biopsy consistent with PBC diagnosis
5. Has documented evidence of cirrhosis and has ALP >ULN and TB ≤5 × ULN

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study:

1. Has consumption of 2 standard alcohol drinks per day (or 14 alcohol drinks per week) if male and 1 standard alcohol drink per day (or 7 alcohol drinks per week) if female for ≥3 consecutive months (12 consecutive weeks) within 5 years prior to screening
2. Has known CPT B (having a score of ≥7) or CPT C (having a score of ≥10) cirrhosis classification at screening
3. Has a Model for End-Stage Liver Disease (MELD)-Na score of ≥12 at screening
4. Has a history or presence of any of the following other concomitant liver diseases at screening:

   i. Chronic hepatitis B or C virus (HBV, HCV) infection. (Note: If a participant has been treated for the HCV infection and has been cured for a duration of >2 years prior to screening, they can be enrolled in the study. Participants who have seroconverted [hepatitis B surface antigen AND hepatitis B antigen is negative] may be included in this study.) ii. Primary sclerosing cholangitis iii. Alcohol-associated liver diseases iv. Autoimmune hepatitis (AIH)-PBC overlap syndrome v. Hemochromatosis vi. Metabolic dysfunction-associated steatohepatitis on historical biopsy vii. α-1 antitrypsin deficiency
5. Has a history or presence of clinically significant hepatic decompensation, including the following:

   i. Liver transplantation or currently placed on a liver transplant list ii. Complications of cirrhosis iii. Hepatorenal syndrome (Type I or II) iv. Known or suspected hepatocellular carcinoma or other hepatobiliary malignancies
6. Use of the following medications (within 12 weeks prior to screening until the randomization [Day 1] visit): thiazolidinediones, fibrates, OCA, methotrexate, budesonide, and other systemic corticosteroids (equivalent to prednisone dose >10 mg); potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazid, and nitrofurantoin); any other newly approved treatments for PBC (eg, elafibranor, seladelpar)
7. Has elevated baseline ALT, AST, or ALP values; ALT, AST, or ALP values increasing by >50% on Visit 2 compared to Visit 1
8. Has any of the following laboratory values:

   i. TB >5 × ULN ii. Platelets <50 × 10^9/L iii. Albumin <2.8 g/dL iv. ALP >10 × ULN v. Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73m^2 vi. ALT or AST >5 × ULN vii. International normalized ratio (INR) >1.7 in the absence of anticoagulant therapy viii. CPK > 2x ULN
9. Has participated in another interventional clinical study and received any other investigational medication or medical device within 30 days or 5 half lives, whichever is longer, prior to screening
10. Has a history of malignancy in the past 5 years and/or active neoplasm, which may diminish life expectancy (except resolved superficial nonmelanoma skin cancer, carcinomas in situ, or other stable, relatively benign conditions prior to screening)
11. Has a known allergy, hypersensitivity, or intolerance to saroglitazar or any of the formulation ingredients
12. Pregnancy-related exclusions, including the following:

    i. If a female, who is pregnant (including a positive pregnancy test at screening), breastfeeding, intends to become pregnant, or is a woman of childbearing potential and not agreeing to use adequate contraceptive methods for at least 1 month after receiving the last dose of the IP ii. Male participants with WOCBP partners and female participants must avoid pregnancy either by true abstinence or the use of acceptable, effective contraceptive measures for the duration of the study and for at least 1 month after receiving the last dose of the IP
13. Has a history or other evidence of severe illness or any other conditions, including cardiovascular, endocrine, hematological, gastrointestinal, neurological, or psychiatric disease, that, in the opinion of the investigator, would make the participant unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of saroglitazar magnesium compared to placebo, based on time to the first occurrence of the defined clinical outcome events in participants with PBC. | baseline to 48 months
  Time from randomization to the first occurrence of any of the following clinical outcome events:
  * Liver decompensation
  * Change in the Model for End-Stage Liver Disease-Na score to ≥15, measured on 2 consecutive occasions, performed at least 2 weeks apart, without the presence of any competing etiologies.
  * Liver transplant.
  * Death (liver- and nonliver-related).
  * Progression to clinically significant portal hypertension, including the variceal related outcomes
  * Progression to Child-Pugh-Turcotte C, defined as Child-Pugh-Turcotte score ≥10, measured at 2 consecutive time points at least 4 weeks apart with no competing etiologies

SECONDARY OUTCOMES:
The incidence of achieving normalization of ALP, defined as ALP ≤ULN | baseline to 12 months
The incidence of achieving normalization of ALP, defined as ALP ≤ULN. | baseline to 48 months
To evaluate the effect of saroglitazar magnesium compared to placebo, based on event-free survival in participants with PBC | baseline to 48 months
  Time from randomization to the first occurrence of any of the following clinical outcome events:
  * Liver decompensation, as defined in the primary endpoint.
  * Liver transplant
  * Death (liver- and non liver-related).
The percentage of participants with stabilization in Total Bilirubin (TB) (ie, no increase), defined as TB ≤1 × ULN or increase from baseline ≤0.1 × ULN | baseline to 48 months
Change from baseline in 'Fatigue Domain Score' of Primary Biliary Cholangitis-40 Quality of Life Questionnaire (PBC-40) | baseline to 12 months
  PBC-40 Fatigue Domain Score consists of 11 question items that measure experience of fatigue over the past week from scale 1 (never) to 5 (always). The PBC-40 Fatigue Domain score ranged from 11 (best) to 55 (worst) (units on a scale). Higher scores indicated worse outcomes. Baseline was defined as the last non-missing value on or before the first dose of the randomized study medication.

IPD SHARING:
Plan to Share IPD: No